CLINICAL TRIAL: NCT01003743
Title: Endolumenal Gastric Pouch and Gastrojejunal Anastomosis Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Other Study IDs: TP165
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Dilated Gastric Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: endolumenal tissue approximation

SUMMARY:
Registry is designed to evaluate use of endolumenal tissue anchors for soft tissue approximation to repair a dilated gastric pouch and gastrojejunal anastomosis in post-Roux-En-Y gastric bypass patients presenting with weight regain. Registry will also assess tissue anchor durability.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age and < 65 years of age
2. Patient is > 2 yrs post-Roux-en-Y bypass surgery
3. Patient initially achieved > 50% EWL after Roux-en-Y bypass surgery
4. Patient is a reasonable risk to undergo general anesthesia
5. Patient is able to provide written informed consent

Exclusion Criteria:

1. Patient has an esophageal stricture or other anatomy/condition that would preclude the use and passage of the endolumenal instruments
2. Physician determines another causal factor for weight regain other than stoma or pouch dilation
3. Patient is non-mobile or has significant impairment of mobility that will limit compliance with post-op exercise

Ages: 19 Years to 64 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States